CLINICAL TRIAL: NCT02672839
Title: A Single-Center, Randomized, Open-Label, 2-Period Complete Crossover Study to Compare the Bioavailability of a Capsule Formulation of LGD-6972 to an Oral Solution Formulation in Healthy Adult Subjects
Brief Title: A Comparison Study of the Bioavailability of a Capsule Formulation of LGD-6972 to an Oral Solution Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: L6972-03
Record Dates: First submitted 2016-01-27; First posted 2016-02-03 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SBE4-beta-cyclodextrin; betadex; RVT-1502

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 1 Treatment A (Experimental): Healthy subjects will receive a single dose orally of LGD-6972 capsules fasted
  Interventions: Drug: LGD-6972 Capsules
- Period 1 Treatment B (Experimental): Healthy subjects will receive a single dose orally of LGD-6972 solution fasted
  Interventions: Drug: LGD-6972 Solution
- Period 2 Treatment A (Experimental): Healthy subjects will receive a single dose orally of LGD-6972 capsules fasted
  Interventions: Drug: LGD-6972 Capsules
- Period 2 Treatment B (Experimental): Healthy subjects will receive a single dose orally of LGD-6972 solution fasted
  Interventions: Drug: LGD-6972 Solution

INTERVENTIONS:
Drug: LGD-6972 Solution — 15 mg of LGD-6972
  Other Names: LGD-6972 Sodium Salt in Captisol ® (betadex [β-cyclodextrin] sulfobutylether sodium, NF)
  Arms: Period 1 Treatment B; Period 2 Treatment B
Drug: LGD-6972 Capsules — 15 mg LGD-6972
  Other Names: LGD-6972 Sodium Salt Capsules
  Arms: Period 1 Treatment A; Period 2 Treatment A

SUMMARY:
The purpose of this study is to compare relative oral bioavailability of a capsule formulation of LGD-6972 to a solution formulation of LGD-6972.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label, single dose study conducted in a 2-way crossover design.

A total of 8 subjects will be enrolled in the study. The duration of participation for each subject will be approximately 36 days, not including a Screening Period of up to 30 days.

Each treatment period, subjects will be admitted to the study site on Day -1 and observed through the morning of Day 3 (48-hour post-dose assessment). Over 2 treatment periods, subjects will receive each of the following treatments as a single dose orally, under fasting conditions, per the randomization (4 subjects per treatment in each treatment period:

Treatment A - 15 mg of LGD-6972 as capsules

Treatment B - 15 mg LGD-6972 as solution

Serial blood samples will be collected through 48 hours following each dose to determine the concentration of LGD 6972 in plasma. Safety assessments will also occur during this time. Subjects will be discharged from the study site after the 48 hour assessments and return to the study site on Days 4, 7, and 14 for follow up procedures. Subjects will return to the study site for the second treatment period after an additional 7 days. Subjects will be discharged from the study after returning to the study site on Day 14 of the second treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult man or woman, 21 to 65 years of age. If the subject is a woman, she must be surgically sterile (hysterectomy or bilateral oophorectomy or bilateral tubal ligation), or naturally post menopausal for at least 12 months and with a follicle stimulating hormone (FSH) level in the post-menopausal range (if not taking hormone replacement therapy) to be considered for enrollment
2. Willing and able to provide written informed consent
3. Not diabetic and has a fasting blood glucose between 70 and 105 mg/dL, inclusive
4. In good health with no significant concomitant pathology based on medical history, physical examination, ECG, routine laboratory tests (chemistry, hematology, lipid profile, and urinalysis), and vital signs
5. Has a body mass index (BMI) between 18.5 kg/m2 and 30 kg/m2, inclusive, and must weigh more than 45 kg
6. Male subjects must either have a vasectomy or agree that they and any female partners will use 2 acceptable forms of contraception, one of which must be a condom, until 30 days after the last dose of study drug. Other acceptable forms of contraception include hormonal contraceptives, intrauterine device, Depo Provera®, Norplant® System Implants, bilateral tubal ligation, bilateral oophorectomy, hysterectomy, and contraceptive sponge, foam, or jelly.

Exclusion Criteria:

1. History of drug and/or alcohol abuse within 2 years prior to screening
2. Unwilling to comply with tobacco, nicotine, alcohol, and caffeine restrictions outlined in the protocol
3. Unwilling to comply with restrictions on strenuous exercise as specified in the protocol
4. Has a history of clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal (including pancreatitis), or metabolic disease requiring medical treatment or has any medical problems that pose an increased risk during the study or that may compromise the integrity of the study data
5. Has liver transaminase levels (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) 10% of the upper limit of normal (ULN), or has creatine kinase (CK) levels 2 × ULN at screening or admission to site (Day 1). Abnormal values at screening may be retested once
6. Has a serum triglyceride level 400 mg/dL at screening. If the triglyceride level is between 400 mg/dL and 500 mg/dL, one retest is permitted
7. Recent history of uncontrolled high blood pressure or has systolic blood pressure 90 mmHg or 140 mmHg or diastolic blood pressure 50 mmHg or 90 mmHg at screening. One or more retests of blood pressure within a reasonable period of time are permissible at the discretion of the Investigator
8. Is taking prescription or non-prescription drugs other than those outlined in the protocol
9. Has a positive screening for hepatitis B virus (HBV), hepatitis C virus (HCV), and/or human immunodeficiency virus (HIV)
10. Woman of childbearing potential
11. Lactating or has a positive pregnancy test
12. Has donated 450 mL of blood within 56 days of admission to the investigational site or has donated blood products within 30 days of admission.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Analysis- Area Under the Concentration Curve (AUC) | Pre-dose, 1,2,4,6,8,10,12,16,24,36,48,72 hrs, 7 and 14 days post dose
  AUC: ratio: medium test form to reference form
Pharmacokinetics Analysis- Maximum Concentration (Cmax) | Pre-dose, 1,2,4,6,8,10,12,16,24,36,48,72 hrs, 7 and 14 days post dose
  Cmax: ratio: medium test form to reference form

SECONDARY OUTCOMES:
Severity of all Adverse Events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) | Day -1, 24, 48, 72hrs, and 7day and 14day post dose
  The severity of all adverse events will be graded according to the CTCAE version 4.0 from dosing until 14 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Biernat, M.D., Principal Investigator — Medpace Clinical Pharmacology
Locations (1):
- Medpace, Inc, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes